CLINICAL TRIAL: NCT06481449
Title: Definitive Radiotherapy for Cervical and Upper Thoracic Esophageal Cancer (ChC&UES): A Multi-center Real World Study
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Fujian Cancer Hospital (Other Government); Fudan University (Other); Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KY155
Record Dates: First submitted 2024-06-22; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High dose radiotherapy (≥60Gy): Patients who received 60 Gy or more than 60Gy radiation dose for radical radiation therapy for the primary tumor.
- Low dose radiotherapy (50-<60Gy): Patients who received 50-<60Gy radiation dose for radical radiation therapy for the primary tumor.

SUMMARY:
Cervical and upper thoracic esophageal cancer (ESCA) presents treatment challenges due to limited clinical evidence. This multi-center study (ChC&UES) explores radical radio(chemo)therapy efficacy and safety

DETAILED DESCRIPTION:
Cervical and upper thoracic esophageal cancer (ESCA) are relatively rare diseases, presenting treatment challenges due to limited clinical evidence. This multi-center study (ChC&UES) explores radical radiotherapy efficacy and safety, especially focusing on radiation dose. This study collected all eligible patients diagnosed with cervical and upper thoracic ESCA from 6 medical centers (Tianjin Cancer Hospital, Cancer Hospital of the Chinese Academy of Medical Sciences, Fujian Cancer Hospital, Fudan University Shanghai Cancer Center, Shandong Cancer Hospital and the Fourth Hospital of Hebei Medical University) in China. Patients were categoried into two group (low dose radiation group and high dose radiation group) based on radiation dose. Basic clinical information, including age, gender, ECOG score, pathological type, smoking and drinking history, initial visit date, radiotherapy dose, radiotherapy method, concurrent chemotherapy modality, immunotherapy, targeted drug usage, treatment efficacy assessment, toxicity and side effects and survival time was collected. Kaplan-Meier method was used to calculate OS, survival differences were assessed using the log-rank test. Univariate analysis was conducted via Cox regression modeling, with variables demonstrating P values < 0.1 being included in multivariate analysis. A significance level of two-sided P < 0.05 was considered statistically significant. The aim of this study was to compared the overall survival time between low dose radiation group and high dose radiation dose group and compared the underlying side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older.
2. Confirmation of esophageal cancer through histopathology or cytology.
3. Primary tumor location within the cervical or upper thoracic segment, extending from the upper esophageal sphincter to the azygos vein.
4. Absence of distant metastasis.
5. Patients unable or unwilling to undergo surgical treatment for various reasons.
6. Receipt of radical radiotherapy as the first-line treatment, with or without chemotherapy, immunotherapy, or targeted therapy.
7. Undergoing conventional radiation therapy (1.8-2.0Gy per session, once per day).
8. Receiving 3DCRT or IMRT radiotherapy.
9. Availability of complete radiotherapy prescription dose information and follow-up records.

Exclusion Criteria:

1. Receipt of radiation dose below 50Gy.
2. History of other malignancies (except for cured cancer in situ and malignancies cured for over 5 years) or laryngeal invasion.
3. Diagnosis of double primary esophageal cancer.
4. Prior chest radiation therapy within the past 5 years.
5. Recurrent or metastatic esophageal cancer.
6. Receipt of 2D radiotherapy, large fractionation, or hyper-fractionation radiotherapy.
7. Patients with incomplete radiotherapy dose and follow-up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a real-world study. All esophageal cancer patients over 18 years old who received radical radiotherapy in cervical and upper thoracic segment eligible for inclusion were retrospectively collected. This study is a reflection of real-world, no restriction on treatment was made.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival time (OS) | 2000.1.1-2024.6.20
  Compared the differences in overall survival (OS) between low dose radiation and high dose radiation group after definitive radiotherapy. OS is defined as time from start of enrollment to death from any cause.
progression-free survival (PFS) | 2000.1.1-2024.6.20
  Progression-free survival (PFS) is defined as the time from the start of enrollment until tumor progression or death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2000.1.1-2024.6.20
  The Objective Response Rate (ORR) is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Measures the effectiveness of a cancer treatment by showing the percentage of patients whose tumors shrink significantly within a specified time. ORR includes: Complete Response (CR): All target tumors disappear, and no new tumors appear.Partial Response (PR): The size of target tumors decreases by at least 30%, and no new tumors appear. The proportion of patients who achieve CR+PR was ORR.

OTHER OUTCOMES:
Side effect | 2000.1.1-2024.6.20
  The investigators employed the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, to assess treatment-related adverse effects during and after the course of treatmen

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Shen, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Because this study is a response to real-world patient treatment and outcomes, Shijiazhuang, Hebei, China